CLINICAL TRIAL: NCT02311205
Title: A Phase II, Prospective, Open-label, Single Arm Study of the Efficacy and Safety of Concurrent Conventional TACE and Sorafenib in Patients With Hepatocellular Carcinoma and Extrahepatic Metastasis (COTSOM Study)
Brief Title: Efficacy and Safety of Concurrent TACE and Sorafenib in Patients With HCC and Extrahepatic Metastasis (COTSOM Study)
Acronym: COTSOM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Kang Mo Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0902
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Hepatocellular Carcinoma; Metastasis
Keywords: Transarterial Chemoembolization (TACE); Hepatocellular carcinoma (HCC); Metastasis; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TACE+sorafenib (Experimental): Concurrent Conventional Transarterial Chemoembolization (TACE) and Sorafenib
  Interventions: Procedure: Conventional Transarterial Chemoembolization (TACE); Drug: sorafenib

INTERVENTIONS:
Procedure: Conventional Transarterial Chemoembolization (TACE) — On demand conventional TACE will be performed in all the patients after enrollment and can be continued until intrahepatic CR, TACE failure or consent withdrawal. Sorafenib will be started 3-7 days after the first and each subsequent TACE and stopped one day before next TACE and will be continued until sorafenib failure, consent withdrawal or condition worsening by clinical decision.
Drug: sorafenib — Sorafenib will be started 3-7 days after the first and each subsequent TACE and stopped one day before next TACE and will be continued until sorafenib failure, consent withdrawal or condition worsening by clinical decision.
  Other Names: nexavar

SUMMARY:
This study is a phase II, prospective, open-label, single arm, single center study of the efficacy and safety of concurrent conventional transarterial chemoembolization (TACE) and sorafenib in patients with hepatocellular carcinoma and extrahepatic metastasis. All of the 55 patients with hepatocellular carcinoma and newly diagnosed extrahepatic (lung, bone, lymph node, adrenal gland) metastasis will be included.

On demand conventional TACE will be performed in all the patients after enrollment and can be continued until intrahepatic CR, TACE failure or consent withdrawal. Sorafenib will be started 3-7 days after the first and each subsequent TACE and stopped one day before next TACE and will be continued until sorafenib failure, consent withdrawal or condition worsening by clinical decision. Repeated on-demand TACE and sorafenib should continue until the criteria for treatment discontinuation are met. After initiation of sorafenib combination treatment, patients will be seen and will perform routine examination at week 4 and, after then routine examination will be followed every 6 ± 2 weeks.

DETAILED DESCRIPTION:
This is a single center, single arm, prospective, phase II study in patients with metastatic HCC. A total of 55 patients with HCC and newly diagnosed extrahepatic (lung, bone, lymph node, adrenal gland) metastasis will be enrolled.

On demand conventional TACE will be performed in all the patients after enrollment and can be continued until intrahepatic CR, TACE failure or consent withdrawal. Safety will be evaluated every 6 ± 2 weeks after initial TACE and closed monitoring at unscheduled visit will be done as well. The efficacy of TACE will be evaluated every 6 ± 2 weeks after each session of TACE using dynamic CT or MRI. Performance of repeated TACE will be decided based on the findings of follow-up CT, patients' liver function and performance status, within 6 ± 2 weeks of the previous TACE. Patients with no residual viable tumors after previous TACE who are not indicated for further TACE are evaluated with routine examination and imaging studies every 6 ± 2 weeks. Safety should be evaluated on an ongoing basis and within 3 days of next TACE. All eligible patients will be given sorafenib (initially 400mg po bid) on day 3-7 after the first or every session of TACE, and sorafenib will be stopped one day before each TACE. Sorafenib will be continued until sorafenib failure, consent withdrawal or condition worsening by clinical decision. Treatment failure will be judged by the evaluation of intra- or extrahepatic lesion separately. TACE failure is defined as when TACE/transarterial chemo-lipiodolization (TACL) has no more benefit by clinical assessment which is judged clinically by one investigator and/or the patient is not more eligible because of worsening of ECOG PS or liver function. Detailed criteria for stopping TACE will be clarified in below. Sorafenib failure will be evaluated by modified RECIST applied to the extrahepatic lesion, and sorafenib will be stopped when progressive disease (PD) by mRECIST for extrahepatic lesion is indicated and clinical benefit of TACE is not expected for intrahepatic lesion. As long as TACE is evaluated to be beneficial and planned to be performed by investigator, sorafenib could be continued if side effect is tolerable.

When any of the treatment discontinuation criteria is met, test treatment will be stopped. Survival and post-treatment information will be collected at 1-3 months intervals after the last study visit until the endpoint of death, or until the subject has become lost to follow-up or until study termination by Principal Investigator. Additional palliative anti-cancer therapies such as cytotoxic chemotherapy and TACL without gelfoam embolization and palliative radiation therapy will be allowed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC and newly diagnosed extrahepatic metastasis meeting of following criteria

  1. Clinical or histological diagnosis of HCC based on the guidelines: Early enhancement followed by late wash-out on dynamic liver imaging (CT or MRI) Or Pathological examination of liver biopsy
  2. Evidence of extrahepatic metastasis with any of following methods; CT, MRI, bone scan, positron emission tomography with FDG-PET, biopsy of metastatic lesion
  3. Preserved liver function classified as Child-Pugh A
  4. ECOG PS of 0-1
  5. Age of at least 20 years
  6. Patients is able to comply with scheduled visits, evaluation plan, and other study procedures
  7. Patient is willing to provide written informed consent
  8. There is no limitation of prior TACE session number in case that further TACE is still considered to be beneficial
  9. Women of childbearing potential must have a negative pregnancy test performed within 14 days of the start of treatment. All patients of child-bearing potential must use adequate birth control measures during the course of the trial (barrier method of birth control) and up to at least 30 days of last dose.

Exclusion Criteria:

* Presence of any of following criteria

  1. Patients who are diagnosed as not eligible for further TACE before screening
  2. Patients with advanced liver disease as defined below:

     * Child Pugh B and C
     * Encephalopathy
     * Ascites
  3. Complete occlusion of main portal vein (PV) by HCC
  4. Patients with brain metastasis
  5. Inadequate liver function that could not perform TACE:

     * AST > 5 X ULN(upper limit normal) or ALT > 5 X ULN
     * Total bilirubin > 2.0 mg/dL
     * Prothrombin time INR > 1.7
  6. Inadequate bone marrow function (absolute neutrophil count < 1,500/μL, Hemoglobin (Hgb) < 8 g/dL, platelet count < 50,000/μL)
  7. Inadequate renal function (creatinine > 1.5 x ULN)
  8. Treatment with previous local therapy such as resection of HCC, radiofrequency ablation (RFA), percutaneous ethanol injection (PEI) < 4 weeks prior to the screening
  9. Prior sorafenib use
  10. Investigational drugs or other molecular target drugs ongoing or completed < 4 weeks prior to the screening
  11. Clinically significant gastrointestinal bleeding within 4 weeks prior to start of study drug
  12. Uncontrolled bleeding varices.
  13. History of cardiac disease:

      * Congestive heart failure >NYHA class 2
      * Active coronary artery disease (CAD) (myocardial infarction more than 6 months prior to study entry is allowed)
      * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before screening
      * Cardiac arrhythmias which are poorly controlled with anti-arrhythmic therapy or requiring pace maker
      * Uncontrolled hypertension
  14. Active clinically serious infections except for HBV and HCV infection
  15. Patients with HIV
  16. Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) within 6 months before screening
  17. Recently treated or concurrent cancer that has a primary site or histology distinct from HCC except any cancer curatively treated more than 3 years prior to screening
  18. Pregnant or breast-feeding subjects
  19. Major surgery, open biopsy, or significant traumatic injury 4 weeks before screening
  20. Presence of a non-healing wound, non-healing ulcer, or bone fracture
  21. Subjects who have used strong CYP3A4 inducers within 4 weeks before screening
  22. Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial
  23. Any other condition which, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the completing the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 1 year from the start of first TACE as a part of combination treatment
  Overall survival (OS) from the start of first TACE as a part of combination treatment

SECONDARY OUTCOMES:
Safety (adverse events and laboratory values) | Up to 1 year from the start of first TACE as a part of combination treatment
  adverse events and laboratory values
Liver dysfunction (laboratory values related to liver) | Up to 1 year from the start of first TACE as a part of combination treatment
  Liver dysfunction (laboratory values related to liver)
Time to progression (TTP) | Up to 1 year from the start of first TACE as a part of combination treatment
Time to TACE failure (TTTF) | Up to 1 year from the start of first TACE as a part of combination treatment
Time to sorafenib failure (TTSF) | Up to 1 year from the start of first TACE as a part of combination treatment
Tumor response rate (TRR) | Up to 1 year from the start of first TACE as a part of combination treatment
  defined as the sum of complete response and partial response, overall, intrahepatic or extrahepatic response respectively
Disease control rate (DCR) | Up to 1 year from the start of first TACE as a part of combination treatment
  defined as the sum of complete response, partial response and stable disease, overall, intrahepatic or extrahepatic response respectively. SD will be decided when it last at least more than 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kang Mo Kim, MD, PhD, Principal Investigator — Asan Medical Center, University of Ulsan
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] Pang RW, Poon RT. From molecular biology to targeted therapies for hepatocellular carcinoma: the future is now. Oncology. 2007;72 Suppl 1:30-44. doi: 10.1159/000111705. Epub 2007 Dec 13. PMID 18087180
- [Background] Kim KM, Kim JH, Park IS, Ko GY, Yoon HK, Sung KB, Lim YS, Lee HC, Chung YH, Lee YS, Suh DJ. Reappraisal of repeated transarterial chemoembolization in the treatment of hepatocellular carcinoma with portal vein invasion. J Gastroenterol Hepatol. 2009 May;24(5):806-14. doi: 10.1111/j.1440-1746.2008.05728.x. Epub 2009 Jan 13. PMID 19207681
- [Background] Kudo M, Izumi N, Kokudo N, Matsui O, Sakamoto M, Nakashima O, Kojiro M, Makuuchi M; HCC Expert Panel of Japan Society of Hepatology. Management of hepatocellular carcinoma in Japan: Consensus-Based Clinical Practice Guidelines proposed by the Japan Society of Hepatology (JSH) 2010 updated version. Dig Dis. 2011;29(3):339-64. doi: 10.1159/000327577. Epub 2011 Aug 9. PMID 21829027
- [Background] Yoo DJ, Kim KM, Jin YJ, Shim JH, Ko GY, Yoon HK, Sung KB, Lee JL, Kang YK, Lim YS, Lee HC, Chung YH, Lee YS, Suh DJ. Clinical outcome of 251 patients with extrahepatic metastasis at initial diagnosis of hepatocellular carcinoma: does transarterial chemoembolization improve survival in these patients? J Gastroenterol Hepatol. 2011 Jan;26(1):145-54. doi: 10.1111/j.1440-1746.2010.06341.x. PMID 21175808
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033